CLINICAL TRIAL: NCT06842979
Title: Effects of Home-based Telerehabilitation-assisted High-intensity Inspiratory Muscle Training on Pelvic Floor Muscle Function and Urinary Symptoms in Women With Stress Urinary Incontinence: A Randomized Controlled Study
Brief Title: Effects of Home-based High-intensity Inspiratory Muscle Training for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Ridvan Aktan, Asst. Prof., PhD, Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023/16-03
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: inspiratory muscle training; stress urinary incontinence; pelvic floor muscle; telerehabilitation
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: This study was designed as a prospective and Randomized Controlled experimental study. Participants were randomly divided into two groups in a 1:1 ratio; the study group and the control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Patients who perform inspiratory muscle training (IMT) with %60 loading
  Interventions: Device: Inspiratory Muscle Training (IMT)
- Sham Group (Sham Comparator): Patients who perform Sham IMT
  Interventions: Device: Sham IMT

INTERVENTIONS:
Device: Inspiratory Muscle Training (IMT) — The IMT protocol will consist of home-based high-intensity daily training - two cycles of 30 breaths with a 1-min rest between sets, twice a day for 8 weeks using an IMT Threshold device (Threshold IMT Philips® Respironics, Inc). The intensity of the training will be set to 60% of each patient's maximal inspiratory pressure measured and adjusted weekly based on the modified Borg scale from 4 to 6 regarding respiratory effort performed during the session. Patients were also informed to perform knack maneuver in daily activities that may cause sudden intra-abdominal pressure overload.
  Arms: Study Group
Device: Sham IMT — The IMT protocol will consist of home-based daily training - two cycles of 30 breaths with a 1-min rest between sets, twice a day for 8 weeks using an IMT Threshold device (Threshold IMT Philips® Respironics, Inc). The intensity of the training will be set to the lowest intensity of the IMT Threshold device. Patients were also informed to perform knack maneuver in daily activities that may cause sudden intra-abdominal pressure overload.
  Arms: Sham Group

SUMMARY:
Strengthening the diaphragm muscle, the roof of the pelvic floor muscles (PFM), may be an alternative intervention in patients suffering from stress urinary incontinence (SUI). This study aims to investigate the effects of home-based telerehabilitation-assisted high-intensity inspiratory muscle training (IMT) on PFM function and urinary symptoms in women with SUI.

DETAILED DESCRIPTION:
The IMT protocol consisted of home-based high-intensity daily training - two cycles of 30 breaths with a 1-minute rest between sets, twice a day for 8 weeks using an IMT Threshold device (Threshold IMT Philips® Respironics, Inc). The IMT was performed twice a day, 7 days/week, for 8 weeks. The study group performed IMT at 60% of their baseline MIP and was adjusted weekly based on the modified Borg scale from 4 to 6 regarding respiratory effort performed during the session, while the control group performed a sham-IMT without applied resistance. Patients are evaluated before the inspiratory muscle training and after 8 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stress urinary incontinence by a specialized Urologist
* Being female aged between 25 and 50 years
* To have the ability to access and use technological devices required by the study
* Being able to read and write
* Volunteering to research

Exclusion Criteria:

* Inability of the participant to understand or perform the procedures proposed during the evaluations or training program.
* Active urinary tract infection,
* pelvic organ prolapse stage 2 and more according to the pelvic organ prolapse staging system (Pelvic Organ Prolapse Quantification System (POP-Q))
* Fecal incontinence,
* Any neurogenic dysfunction of the lower urinary tract
* Conservative or surgical treatment of urinary incontinence in the last 12 months
* Previous pelvic floor training
* Less than three months after pregnancy or postpartum
* Having undergone any pelvic floor surgery (hysterectomy, etc.)
* Radiotherapy treatment in the last 12 months
* Severe low back pain or pelvic pain
* Lower extremity orthopaedic problems that may affect the pelvic structure (such as lower extremity inequality, total hip arthroplasty)
* Having any chronic respiratory disease
* Having any neurological disease
* Being in menopause
* Latex allergy

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Change of Pelvic floor muscle functions with Pressure feedbacks | 8 weeks
  Pressure feedbacks: Pelvic muscle functions were evaluated with pressure feedback of pelvic muscle using a biofeedback device (Myomed 932®- Enraf-Nonius, Delf, The Netherlands), and recorded in hPa (Hectopascal).
  - Manual muscle test: Manual muscle test was evaluated using the modified Oxford Scale that ranges from 1 to 5. Higher values on this scale indicate better muscle strength.
Change of Pelvic floor muscle functions with Manual muscle test | 8 weeks
  The manual muscle test was evaluated using the modified Oxford Scale, which ranges from 1 to 5. Higher values on this scale indicate better muscle strength.

SECONDARY OUTCOMES:
Urogenital Distress Inventory-Short Form | 8 weeks
  Urinary symptom was assessed with the Urogenital Distress Inventory-Short Form (range: 0-100) Higher values on this scale indicate worse symptoms.
International Consultation on Incontinence Questionnaire-Short Form | 8 weeks
  Urinary incontinence symptom and its effect on the quality of life was assessed with the International Consultation on Incontinence Questionnaire-Short Form (range: 0-21) Higher values on this scale indicate worse symptoms.
Incontinence Severity Index | 8 weeks
  Urinary incontinence severity was assessed with the Incontinence Severity Index (range: 1-12). Higher values on this scale indicate worse symptoms.
Inspiratory muscle strength | 8 weeks
  The Inspiratory muscle strength was evaluated by maximum inspiratory pressure which was assessed with a digital mouth pressure meter device (MicroRPM, Micro Medical Ltd., Rochester, Kent, United Kingdom), and recorded in cmH2O (centimeter-water).

CONTACTS AND LOCATIONS:
Overall Officials: RIDVAN AKTAN, Asst. Prof., Principal Investigator — Izmir University of Economics
Locations (1):
- Izmir University of Economics, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Hodges PW, Gandevia SC. Changes in intra-abdominal pressure during postural and respiratory activation of the human diaphragm. J Appl Physiol (1985). 2000 Sep;89(3):967-76. doi: 10.1152/jappl.2000.89.3.967. PMID 10956340
- [Background] Talasz H, Kofler M, Kalchschmid E, Pretterklieber M, Lechleitner M. Breathing with the pelvic floor? Correlation of pelvic floor muscle function and expiratory flows in healthy young nulliparous women. Int Urogynecol J. 2010 Apr;21(4):475-81. doi: 10.1007/s00192-009-1060-1. Epub 2009 Dec 8. PMID 19997721
- [Background] Talasz H, Kremser C, Kofler M, Kalchschmid E, Lechleitner M, Rudisch A. Phase-locked parallel movement of diaphragm and pelvic floor during breathing and coughing-a dynamic MRI investigation in healthy females. Int Urogynecol J. 2011 Jan;22(1):61-8. doi: 10.1007/s00192-010-1240-z. Epub 2010 Aug 31. PMID 20809211
- [Background] Al-Bilbeisi F, McCOOL FD. Diaphragm recruitment during nonrespiratory activities. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):456-9. doi: 10.1164/ajrccm.162.2.9908059. PMID 10934070
- [Background] CAMPBELL EJ, GREEN JH. The variations in intra-abdominal pressure and the activity of the abdominal muscles during breathing; a study in man. J Physiol. 1953 Nov 28;122(2):282-90. doi: 10.1113/jphysiol.1953.sp004999. No abstract available. PMID 13118539
- [Background] Neumann P, Gill V. Pelvic floor and abdominal muscle interaction: EMG activity and intra-abdominal pressure. Int Urogynecol J Pelvic Floor Dysfunct. 2002;13(2):125-32. doi: 10.1007/s001920200027. PMID 12054180
- [Background] Sapsford RR, Hodges PW, Richardson CA, Cooper DH, Markwell SJ, Jull GA. Co-activation of the abdominal and pelvic floor muscles during voluntary exercises. Neurourol Urodyn. 2001;20(1):31-42. doi: 10.1002/1520-6777(2001)20:13.0.co;2-p. PMID 11135380
- [Background] Saunders SW, Rath D, Hodges PW. Postural and respiratory activation of the trunk muscles changes with mode and speed of locomotion. Gait Posture. 2004 Dec;20(3):280-90. doi: 10.1016/j.gaitpost.2003.10.003. PMID 15531175
- [Background] Azevedo IG, Sousa SLO, Viana ESR, Dantas DS, Maciel ACC, Da Camara SMA. Relationship between symptomatic pelvic organ prolapse and respiratory muscle strength in middle-aged and older women in Northeast Brazil: a cross-sectional study. Physiother Theory Pract. 2021 Jun;37(6):755-761. doi: 10.1080/09593985.2019.1642428. Epub 2019 Jul 11. PMID 31294670
- [Background] Hodges PW, Sapsford R, Pengel LH. Postural and respiratory functions of the pelvic floor muscles. Neurourol Urodyn. 2007;26(3):362-71. doi: 10.1002/nau.20232. PMID 17304528
- [Background] Deffieux X, Hubeaux K, Porcher R, Ismael SS, Raibaut P, Amarenco G. Pelvic floor muscle activity during coughing: altered pattern in women with stress urinary incontinence. Urology. 2007 Sep;70(3):443-7; discussion 447-8. doi: 10.1016/j.urology.2007.03.084. PMID 17905093